CLINICAL TRIAL: NCT04075578
Title: Evaluation of Professional Practices in Botulinum Toxin Type A Intradetrusor Injection, at the Dose of 50 Units for the Treatment of Urinary Incontinence by Refractory Idiopathic Overactive Bladder
Brief Title: Evaluation of Professional Practices in the Treatment of Refractory Idiopathic Overactive Bladder at the Dose of 50 Units (TOX50IUU)
Acronym: TOX50IUU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2019 CAMPAGNE-LOISEAU; 2019-A01296-51 (Other: ANSM)
Record Dates: First submitted 2019-08-29; First posted 2019-08-30 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Bladder, Overactive
Keywords: idiopathic overactive bladder; Botox; Onabotulinum toxinA; 50 units
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- female with urinary incontinence: Female ≥ 18 years, suffers from urinary incontinence by idiopathic overactive bladder, inadequately treated by 2 anticholinergic medicines during a period of 3 months for each of them or stopped for intolerance or adverse events
  Interventions: Drug: OnabotulinumtoxinA / Botox®, Allergan Ltd, Irvine, CA, United-States

INTERVENTIONS:
Drug: OnabotulinumtoxinA / Botox®, Allergan Ltd, Irvine, CA, United-States — Botox® intradetrusor injections, with a rigid cystoscope, under local anaesthesia performed by Lidocaïne 2% diluted in 30ml of bicarbonate 14‰. 20 injections of 0,5ml each will be heterogeneously administrated into the bladder wall, sparing the trigone

SUMMARY:
Considering that the 2013 Hermieu's guidelines differs from the product marketing authorization delivered in November 2014, the primary endpoints is to evaluate life quality by questionnaires at the baseline time, and after two, six and twelve weeks of treatment in patients suffer from urinary incontinence by refractory idiopathic overactive bladder and treated by Botox® at the dose of 50UI (international units)

DETAILED DESCRIPTION:
Currently, Botox injection is one of the second-line treatments for urinary incontinence by idiopathic overactive bladder. Multiple studies have shown that Botox at the dose of 50UI is effective but not for a long time. Maximum efficiency is about two weeks and until about twelve weeks compared to the dose between 100UI and 300UI that shown an efficiency until twenty-four at thirty-six weeks. But it's not without consequence since the side effects are more numerous increasing the dose. The most frequent are urinary retention with necessary to perform clean intermittent catheterization and urinary infection.

This dose at 50UI is therefore more a test to assess the patient's tolerance to the product, as recommended by the product marketing authorization.

So, through this evaluation of professional practices, investigators would like to evaluate the patient satisfaction treated in hospital, with a first dose at 50UI.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age ≥ 18 yo
* Refractory idiopathic overactive bladder
* Eligibility to an injection treatment
* Capacity to perform clean intermittent catheterization

Exclusion Criteria:

* Protected adults (under trusteeship, guardianship or judicial protection)
* Patients under anticholinergics for an other desease (psychiatric, neurologic for example)
* Known hypersensitivity or at risk of hypersensitivity to botulinum toxin type A like myasthenic syndrom
* Patients who suffer from an overactive bladder with a known cause (neurological, urological condition)
* urinary infection under treatment < 48 hours before Botox® injections
* Suspicious looking bladder requiring biopsies during the cystoscopy
* Pregnant or breastfeeding women
* Language barriers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female ≥ 18 yo, suffers from urinary incontinence by idiopathic overactive bladder, inadequately treated by 2 anticholinergic medicines during a period of 3 months for each of them or stopped for intolerance or adverse events
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-06-26 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the life quality by the KHQ (King's Health Questionnaire) | Week 6
  Patients will have to answer the questionnaire at home depending the symptoms that they feel at 6 weeks. The data will then be collected by phone

SECONDARY OUTCOMES:
Evaluation of the life quality by the USP (Urinary Symptom Profile) questionnaire | Week 2
  Patients will have to answer the questionnaires at home depending the symptoms that they feel. The data will then be collected by phone. The data will then be collected and analysed.
Evaluation of the life quality by the USP (Urinary Symptom Profile) questionnaire | Week 12
  Patients will have to answer the questionnaires at home depending the symptoms that they feel. The data will then be collected during the postoperative consultation. The data will then be collected and analysed.
Evaluation of the life quality by the KHQ (King's Health Questionnaire) | Week 2
  Patients will have to answer the questionnaires at home depending the symptoms that they feel. The data will then be collected by phone at 2 weeks. The data will then be collected and analysed
Evaluation of the life quality by the KHQ (King's Health Questionnaire) | Week 12
  Patients will have to answer the questionnaires at home depending the symptoms that they feel. The data will then be collected during the postoperative consultation. The data will then be collected and analysed
Patient experience's evaluation of the local anaesthesia and outpatient care thanks to the EVAN-LR (Evaluation du Vécu de l'ANesthésie Loco-Régionale) questionnaire | Day 1
  Patients will have to answer the questionnaire before the return home just after the injection session to assess their experience concerning local anaesthesia and outpatient management.

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine CAMPAGNE-LOISEAU, PH, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France